CLINICAL TRIAL: NCT00554580
Title: Effect of Continuous Positive Airway Pressure on Short Term Inhospital Prognosis for Acute Pulmonary Edema
Brief Title: Continuous Positive Airway Pressure for Acute Pulmonary Edema
Acronym: CPAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem TOUHAMI-CARRIER, Department clinical research of the developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 030428; AOM 03073
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Pulmonary Edema; Dyspnea; Paroxysmal; Congestive Heart Failure
Keywords: continuous positive airway pressure; outcome measure; clinical trial
MeSH Terms: conditions — Pulmonary Edema; Dyspnea; Heart Failure | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Usual care of pulmonary acute oedema
  Interventions: Procedure: usual care of acute pulmonary oedema
- B (Experimental): CPAP + usual care of pulmonary acute oedema
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure (CPAP) — Usual treatment of acute pulmonary oedema (see arm A) + CPAP will be administered without interruption for at least one hour and will be stopped for efficacy:
  stade I or II KILLIP classification and FR less or equal to 25 /min and SpO2 larger than 90 % ambient air and patient willing the stop of CPAP because of improvement of his clinical status.
  Arms: B
Procedure: usual care of acute pulmonary oedema — Usual treatment of acute pulmonary oedema including :
  Oxygen, diuretic minimum one bolus IV of 40 mg FUROSEMIDE (LASILIX) possibility to repeat the dose every 15 minutes with a maximum 120 mg.
  Bolus of ISOSORBIDE DINITRATE (RISORDAN) of 1 mg maybe repeated every 3 minutes.
  As soon as possible perfusion of ISDN with flow adapted to the clinical status If necessary administration of DOBUTAMINE continuous perfusion of to 5 to 20 µg/kg/min.
  Arms: A

SUMMARY:
The investigators hypothesise that CPAP + pharmaceutical treatment, compared to pharmaceutical treatment alone, improves the respiratory and hemodynamic status of the patients before H2 after the inclusion time and decreases the rate of death and tracheal intubation during the first 48 hours.

DETAILED DESCRIPTION:
Patients are included at home after informed consent by the emergency medical team and transported during the following 2 hours to a cardiac intensive care unit were the treatment is purchased as well. Randomization process has been done previously with envelopes ; group A : pharmaceutical treatment alone , B pharmaceutical plus CPAP. Medical treatment includes furosemide and nitroglycerin (continuous perfusion and bolus), inotropes if needed, and all other specific treatment required (ex : anti antiarrhythmic drugs). Doses are free, adapted to the clinical response for respiratory and hemodynamic distress. CPAP is a passive high flow venturi system device alimented by a hyperbaric oxygen. FiO2 can be controlled and adapted to the pulsed oxygen saturation. PEP must be initially celled at least at 7.5 cmH2O and increased to 10 if well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* acute respiratory insufficiency with hypoxia in air
* KILLIP score from 2 to 4
* absence of known ST elevation acute coronary syndrome
* accepted inform consent.

Exclusion Criteria:

* age < 18
* immediate intubation criteria (bradypnea, coma status)
* refractory shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2004-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Composite criteria includes during the first 48 hours : death, tracheal intubation and mechanical ventilation rates, persistence of inclusion criteria for respiratory distress and shock until H2, reappearance of inclusion criteria after H2. | 48 hours

SECONDARY OUTCOMES:
brain natriuretic factor value curves from H0, H6 and H24; composite criteria without intubation rate; clinical and biological parameters evolution during the first 48 hours, myocardial infarction rate, CPAP non tol | H0, H6, H24, H48

CONTACTS AND LOCATIONS:
Overall Officials: DUCROS Laurent, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- DUCROS Laurent, Paris, France

REFERENCES:
- [Derived] Ducros L, Logeart D, Vicaut E, Henry P, Plaisance P, Collet JP, Broche C, Gueye P, Vergne M, Goetgheber D, Pennec PY, Belpomme V, Tartiere JM, Lagarde S, Placente M, Fievet ML, Montalescot G, Payen D; CPAP collaborative study group. CPAP for acute cardiogenic pulmonary oedema from out-of-hospital to cardiac intensive care unit: a randomised multicentre study. Intensive Care Med. 2011 Sep;37(9):1501-9. doi: 10.1007/s00134-011-2311-4. Epub 2011 Jul 30. PMID 21805159